CLINICAL TRIAL: NCT07371169
Title: Efficacy of Chromium Picolinate in Reducing Acanthosis Nigricans Severity in Adolescents With Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uruk University (Other)
Responsible Party: Principal Investigator, Ghasak kais Abdulhussain, Lecturer in department of Pharmacology (B.Sc , M.Sc, Ph.D) / College of Pharmacy, Uruk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UU-CR-2025-01
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Insulin Resistance; Acanthosis Nigricans
Keywords: Chromium Picolinate; Insulin resistance; Acanthosis Nigricans
MeSH Terms: conditions — Insulin Resistance; Acanthosis Nigricans | interventions — picolinic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a double-blind study. Participants, and outcome assessors, (Physician and laboratory personnel) will be unaware of treatment assignment. Clinical assessment of acanthosis nigricans severity using the Burke quantitative scale for acanthosis nigricans severity and laboratory assessment of insulin resistance using the homeostasis model assessment of insulin resistance, based on fasting plasma glucose and fasting serum insulin measurements, will be performed without knowledge of treatment allocation. The study medication and placebo will be identical in appearance and packaging. Treatment allocation codes will be securely stored and will be revealed only after completion of data analysis, unless unblinding is required for participant safety.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chromium Picolinate (Experimental): Participants in this arm (n=45) will recieve oral Chromium Picolinate 200mcg capsules once daily during the 24-weeks study period.
  Interventions: Drug: Chromium picolinate
- Placebo Control (Placebo Comparator): Participants in this arm (n=45) will recieve oral placebo capsules matching the shape size and color of Chromium Picolinate, once daily during the 24-weeks study period; they will act as the control group.
  Interventions: Drug: Placebo matching Chromium Picolinate

INTERVENTIONS:
Drug: Chromium picolinate — Chromium Picolinate Cap. 200mcg once daily for 24-weeks.
  Arms: Chromium Picolinate
Drug: Placebo matching Chromium Picolinate — An inert capsule identical in appearance and packaging to the chromium picolinate 200 microgram capsule (same size, shape, color, weight, and dosing schedule), manufactured without active ingredient. The capsule shell is composed of gelatin or hypromellose, matching the active capsules. The capsule is filled with inert excipients suitable for oral capsules, such as microcrystalline cellulose and magnesium stearate, to replicate the weight and flow properties of the active capsules. Optional coloring agents are included as needed to match the active product. Capsules are packaged in sealed blisters to minimize odor, taste, and visual cues. Dispensed by the investigational pharmacy according to the randomization schedule; to be taken once daily.
  Arms: Placebo Control

SUMMARY:
The goal of this clinical trial is to learn if chromium picolinate can reduce the severity of acanthosis nigricans and improve insulin resistance in adolescents with both conditions. It will also learn about the safety of chromium picolinate use in this age group. The main questions it aims to answer are:

1. Does chromium picolinate reduce the severity of acanthosis nigricans as measured by the Burke quantitative scale for acanthosis nigricans severity in adolescents with insulin resistance?
2. Does chromium picolinate improve insulin resistance as measured by the homeostasis model assessment of insulin resistance (HOMA-IR)?
3. What medical problems do participants have when taking chromium picolinate? Researchers will compare chromium picolinate to placebo to see if chromium picolinate is effective in reducing acanthosis nigricans severity and improving insulin resistance.

Participants will:

1. Take chromium picolinate or placebo daily for 24 weeks.
2. Acquire baseline assessment and then visit the clinic at 8 weeks, 16 weeks, and 24 weeks for clinical evaluation, acanthosis nigricans severity assessment using the Burke quantitative scale for acanthosis nigricans severity, laboratory assessment of insulin resistance using the homeostasis model assessment of insulin resistance, and monitoring for any side effects or complications.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent patients of both sexes, aged 12 to 18 years.
* Clinically diagnosed with acanthosis nigricans.
* Present Insulin resistance, defined as Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) ≥ 2.5.
* Willing to participate in the study, with written informed consent provided by both the patient and guardian.

Exclusion Criteria:

* Diagnosis of type 1 or type 2 diabetes mellitus.
* Known hypersensitivity to chromium or any of the capsule excipients.
* Use of insulin-sensitizing medications (e.g., metformin, thiazolidinediones) within 3 months before screening.
* Use of systemic corticosteroids or other medications known to affect glucose metabolism within 3 months before screening.
* Significant renal disease (estimated glomerular filtration rate < 60 mL/min/1.73 m²) or liver disease (alanine aminotransferase or aspartate aminotransferase > 2.5 times the upper limit of normal).
* Pregnancy or lactation.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Change in the clinical severity of Acanthosis Nigricans | Baseline, 8 weeks, 16 weeks, 24 weeks from enrollment
  Acanthosis nigricans clinical severity will be measured using the Burke's quantitative scale by a trained physician. The primary outcome is the difference in acanthosis nigricans severity between the chromium picolinate group and the placebo control group.
Change in the severity of insulin resistance | Baseline, 8 weeks, 16 weeks, 24 weeks
  The severity of insulin resistance will be measured using the Homeostasis Model Assessment of Insulin Resistance (HOMA-IR), this involves taking a fasting blood sample to measure plasma glucose and serum insulin and applying the formula (HOMA-IR = (Fasting insulin [µIU/mL] × Fasting glucose [mg/dL]) / 405). The primary outcome is the difference in insulin resistance severity based on HOMA-IR results between the chromium picolinate group and the placebo control group.

CONTACTS AND LOCATIONS:
Overall Officials: Ghasak Kais Abdulhussain, BSc, MSc, PhD (Pharmacology), Principal Investigator — Uruk University
Locations (1):
- Baghdad Medical City / Children Welfare Teaching Hospital / Department of Endocrinology, Baghdad, Baghdad Governorate, Iraq

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data, including acanthosis nigricans severity measurements, insulin resistance severity status, baseline demographics, and follow-up data relevant to primary outcomes.
Time Frame: Upon publication of the trial result on open access repository.
Access Criteria: Access will be open to researchers and the public via a free, open-access data repository, with a DOI provided in the publication. Data will be de-identified to protect participant privacy.
URL: https://www.zenodo.org